CLINICAL TRIAL: NCT04313686
Title: Mindfulness-based Intervention to Promote Psychological Wellbeing in People With Epilepsy: A Randomized Controlled Trial
Brief Title: Mindfulness-based Intervention to Promote Psychological Wellbeing in People With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Professor Dr Lim Kheng Seang, Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20175295282
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Epilepsy; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
Keywords: Mindfulness; Epilepsy; Quality of life; Depression; Psychotherapy
MeSH Terms: conditions — Epilepsy; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based therapy (Experimental): The mindfulness training program included mindfulness meditation practices, self-enquiries, mindful movement as well as understanding of stress physiology and cognitive awareness in the Breathworks/ Paradigm system of mindfulness-based approaches. Participants were enrolled in 5-10-person groups that met weekly for 2-3-hour long sessions for six weeks at the patient's usual follow-up clinic.
  Interventions: Behavioral: Mindfulness-based therapy
- No-Intervention (Active Comparator): The control group would attend their routine follow-up visits at the neurology outpatient clinic.
  Interventions: Behavioral: No-intervention

INTERVENTIONS:
Behavioral: Mindfulness-based therapy — Based on randomization, those who first receive the mindfulness training program are the intervention group. Participants would meet weekly for 2-3-hour long sessions for six weeks at the patient's usual follow-up clinic.
  Arms: Mindfulness-based therapy
Behavioral: No-intervention — Participants who were randomized into this group would continue to receive their usual follow-up care at the usual neurology outpatient clinic.
  Arms: No-Intervention

SUMMARY:
The efficacy of mindfulness-based intervention (MBI) for epilepsy has yet to be thoroughly investigated. Hence, the aim of the present study is to examine the effects of MBI on the psychological wellbeing of people with epilepsy (PWE) using a randomized trial design. Key outcomes include depression, anxiety and quality of life. Our primary objective was to evaluate the effect of mindfulness-based therapy on anxiety, depression, epilepsy specific QOL, and life satisfaction in PWE, applying the concept of Reliable Change Index. The secondary objective was to assess whether the results correlate with the level of mindfulness. Study results may be used to decide whether it is worth offering mindfulness training for PWE as an alternative therapy to cope and improve seizure management.

DETAILED DESCRIPTION:
Epilepsy is a debilitating condition characterized by sudden recurrent episodes of epileptic seizures. Psychiatric comorbidities are common in people with epilepsy (PWE), and the presence is associated with increased rates of suicide, healthcare costs, mortality and reduced quality of life. Studies showed that poor health-related quality of life (HRQOL) has been linked to seizure frequency, medication side effects, psychological disturbances and psychosocial difficulties. Medical therapies aside, psychological interventions like mindfulness-based interventions (MBIs) were proven effective in improving psychological health as well as seizure control. Recent review was conducted to determine the efficacy of MBIs for PWE. Although promising results showed reduction in levels of psychological distress and improvement in quality of life, the extracted findings were based on three articles which limit the applicability of the findings. More research focusing on MBIs for PWE are required to make comparisons on its beneficial effects. Hence, this present study aimed to examine the effects of MBI on psychological wellbeing among PWE using a randomized controlled trial design.

This study trial recruits 30 participants with epilepsy. Participants are recruited from the neurology outpatient treatment clinic and those who consented are randomized into either the intervention active or no-intervention group. All participants receive six weekly-sessions of mindfulness training that lasted for 2.5-hour. Assessments are conducted at three time-points (T0: before intervention, T1: immediately after intervention, and T2: at the 6-weeks followup). The following outcome measures assessing depression (BDI-II), anxiety (BAI), quality of life (QOLIE-31), mindfulness (MAAS) and satisfaction with life (SWLS) are collected at all three time-points.

ELIGIBILITY:
Inclusion Criteria:

* All patients (16 years or older) with a diagnosis of epilepsy by a neurologist and who were able to read and write English.

Exclusion Criteria:

* a diagnosis of severe learning disability or cognitive impairment that affects individuals who are unable to comply with study procedure, substance dependence, suicidality, and limited language proficiency.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Three time-points: T0: (prior to therapy), T1: (immediately after intervention), T2 (three-month after phase one after no-intervention wash-out period)
  Total 21 items measuring cognitive, somatic and affective symptoms of anxiety. Each item is rated on a 4-point Likert scale for symptom severity experienced, ranging from 0 (not at all) to 3 (severely). The scores ranged between 0 to 63, with higher numbers suggesting greater degrees of anxiety.
Beck Depression Inventory (BDI-II) | Three time-points: T0: (prior to therapy), T1: (immediately after intervention), T2 (three-month after phase one after no-intervention wash-out period)
  Total 21 items assessing the presence and severity of depressive symptoms. All descriptive items were scored on a 4-point Likert scale ranging from 0 to 3. Total scores ranged from 0 to 63, higher scores represent higher degrees of depressive symptoms.
Quality of Life in Epilepsy Inventory (QOLIE-31) | Three time-points: T0: (prior to therapy), T1: (immediately after intervention), T2 (three-month after phase one after no-intervention wash-out period)
  Total 31 items reflects the patient's subjective well-being toward his or her QOL in various aspects related to epilepsy, with higher scores indicating better well-being.

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale (MAAS) | Three time-points: T0: (prior to therapy), T1: (immediately after intervention), T2 (three-month after phase one after no-intervention wash-out period)
  Total 15 items were each rated on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never) to measure the core characteristic of dispositional mindfulness.
Satisfaction with Life Scale (SWLS) | Three time-points: T0: (prior to therapy), T1: (immediately after intervention), T2 (three-month after phase one after no-intervention wash-out period)
  Total 5 items were each rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree) to assess one's global cognitive judgements of individual's life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Lim Kheng Seang, MBBS, PhD, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia